CLINICAL TRIAL: NCT04002947
Title: A Phase 2 Study of Acalabrutinib With DA-EPOCH-R or R-CHOP for Patients With Untreated Diffuse Large B-cell Lymphoma
Brief Title: Acalabrutinib With DA-EPOCH-R or R-CHOP for People With Untreated Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190116; 19-C-0116
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12-29

CONDITIONS: Non-Hodgkin's Lymphoma; Diffuse Large B-Cell Lymphoma; DLBCL; NHL
Keywords: BTK Inhibitor; Calquence; ACP-196; Monoclonal Antibody
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — EPOCH protocol; Rituximab; acalabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Acalabrutinib 100 mg orally twice a day for 14 days; Following window: patients with > or = to 25% tumor reduction, treat with DA-EPOCH-R or R-CHOP + acalabrutinib 100mg orally twice a day for the first 10 days, for 6 cycles; whereas, patients with <25% tumor reduction, treat with DA-EPOCH-R or R-CHOP alone for 6 cycles
  Interventions: Drug: DA-EPOCH; Biological: Rituximab; Drug: CHOP; Drug: Acalabrutinib

INTERVENTIONS:
Drug: DA-EPOCH — Vincristine 1.4 mg/m2 (2 mg cap) IV on Day 1, Doxorubicin 10 mg/m2/day CIVI on Days 1-4, Etoposide 50 mg/m2/day CIVI on Days 1-4, Cyclophosphamide 750 mg/m2 IV on Day 5. Prednisone 60 mg/m2 PO BID is administered daily on Days 1-5 of each cycle. Each cycle is 21 days and drugs will be given for 6 cycles.
Biological: Rituximab — Rituximab 375 mg/m2 IV on Day 1 of each 21-day cycle for 6 cycles.
Drug: CHOP — Cyclophosphamide 750 mg/m2 IV, Doxorubicin 50 mg/m2 IV, Vincristine 1.4 mg/m2 (2 mg cap) IV are administered on Day 1 of each 21-day cycle for 6 cycles. Prednisone 40 mg/m2 PO is administered daily on Days 1-5 of each cycle.
Drug: Acalabrutinib — Acalabrutinib is administered orally at 100 mg twice a day for 14 days during the window period. During combination therapy, acalabrutinib is administered 100 mg twice daily for the first 10 days for 6 cycles.

SUMMARY:
Background:

Diffuse large B-cell lymphoma is the most common type of non-Hodgkin lymphoma. Most people with this cancer can be cured. But those who are not cured have a poor prognosis. Researchers want to add another drug to standard treatment see if it can improve the cure rate.

Objective:

To see if the drug acalabrutinib given with rituximab and standard combination chemotherapy can improve the cure rate of aggressive B-cell lymphomas such as diffuse large B-cell lymphoma.

Eligibility:

People ages 18 and older with an aggressive B-cell lymphomas that have not been treated

Design:

Participants will be screened with:

Blood and urine tests

Physical exam

Medical history

Tumor biopsy

Bone marrow biopsy: A needle will remove marrow from the participant s hipbone.

Lumbar puncture: If necessary, a needle will remove fluid from the participant s spinal canal.

Imaging scans

Participants will take the study drug for up to 14 days. It is a pill taken 2 times a day. Then they will have more scans. They will get rituximab and chemotherapy. They may get these drugs through a needle in an arm vein. Or they may them through a tube placed in a vein in their chest or in their neck. They might also keep taking the study drug. Each treatment cycle lasts 21 days. They will have up to 6 cycles.

Participants may have 4 doses of another drug injected into their spinal fluid.

Participants will have repeats of the screening tests throughout the study.

Participants will have a follow-up visit 30 days after their last treatment, then every 3 months for 2 years, then every 6 months for 3 years, and then yearly.

DETAILED DESCRIPTION:
Background:

Gene-expression profiling (GEP) has identified two dominant molecular subtypes, activated B cell like (ABC) and germinal center B cell like (GCB), that arise by distinct mechanisms, have distinct prognoses, and respond differently to targeted therapy

Recently, genetic subtypes of DLBCL have been described within molecular subtypes that have distinct genotypic, epigenetic, and clinical characteristics providing biologic rationale for precision medicine strategies in DLBCL

Frontline treatment of DLBCL is either rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP), or infusional rituximab, cyclophosphamide, doxorubicin, etoposide, vincristine, and prednisone (DA-EPOCH-R) but up to 40% of patients are not cured with frontline treatment

Bruton s tyrosine kinase (BTK) is a key component of the B-cell receptor (BCR)-signaling cascade and selective BTK inhibitors have clinical activity preferentially in ABC-DLBCL

Acalabrutinib is a selective, small molecule, next-generation BTK inhibitor approved for relapsed mantle cell lymphoma and demonstrated activity in DLBCL

The molecular characterization of tumors that respond to DLBCL BTK inhibitors is incomplete; although responses occur more commonly in ABC-DLBCL, cases of GCB-DLBCL show minor responses, and no information is available within genetic subtypes of DLBCL

Patients with minor responses during 2-week window of treatment with acalabrutinib (100mg BID) as a single agent may benefit from acalabrutinib added to standard combination therapy as part of frontline therapy

Objectives:

To determine the response rate, including minor response (MR), to acalabrutinib administered for 14 days in molecular and genetic subtypes of untreated DLBLC (ABC, GCB, unclassified, genetic subtypes)

Eligibility:

Histologically confirmed DLBCL or high-grade B-cell lymphoma

Primary mediastinal B-cell lymphoma (PMBL) and CNS involvement excluded

Stages II-IV

HIV negative or positive

Available FFPE or fresh frozen biopsy

Adequate organ function

Age >= 18 years

Design:

Open-label, single center, non-randomized phase 2 study, with enrollment of 100 untreated DLBCL patients. It is estimated that there may be 50% who are ABC (~50 patients), and 50% who are GCB or unclassified (~50 patients). The accrual ceiling will be set at 132 to allow for inevaluable patients and to account for screen fails.

The study will start with an initial 2-week window of treatment with acalabrutinib (100mg BID) as a single agent, with collection and assessment of molecular correlates as well as response rates (by imaging) by molecular subtype

Treatment with chemoimmunotherapy (R-CHOP or DA-EPOCH-R) either alone or in combination with acalabrutinib will depend on response during window; those with less than 25% reduction during window will receive chemoimmunotherapy alone, while those with at least a 25% reduction in tumor lesions (sum of the products of the longest diameter) will receive combination therapy of chemoimmunotherapy with acalabrutinib (100mg BID on days 1-10 of each cycle); those with clinical progression during window will move immediately to chemoimmunotherapy

Secondary objectives include: integrative genomic analysis of all untreated DLBCL that respond or are resistant to acalabrutinib for 14 days, event-free survival (EFS), assessment of progression free survival (PFS) and overall survival (OS) of combination therapy of

acalabrutinib and chemoimmunotherapy and investigation of the safety and tolerability of acalabrutinib added to R-CHOP or DA-EPOCH-R in untreated DLBCL.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must have a confirmed histologic diagnosis of an aggressive B-cell lymphoma with morphologic appearance of DLBCL or high-grade B-cell lymphoma (HGBL) confirmed by the Laboratory of Pathology, NCI, with no prior treatment for DLBCL or HGBL. The following subtypes are included:

   * DLBCL, NOS, Activated B-cell type (ABC)
   * DLBCL, NOS, Germinal center B-cell type (GCB)
   * T-cell/histiocyte-rich large B-cell lymphoma
   * Primary cutaneous DLBCL, leg-type
   * EBV+ DLBCL, NOS
   * DLBCL associated with chronic inflammation
   * ALK+ large B-cell lymphoma
   * High-grade B-cell lymphoma, NOS
   * High-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements

   NOTE: Presence of concomitant indolent lymphomas such as follicular lymphoma, marginal zone lymphomas, monoclonal B-cell lymphocytosis or chronic lymphocytic leukemia/small lymphocytic lymphoma that are best categorized as composite or transformed lymphomas are allowed.
2. A formalin-fixed tissue block or 15 slide of tumor sample (archival or fresh) must be available for performance of correlative studies.

   NOTE: Tumor tissue may be from any previously collected tissue and adequacy is at the discretion of the Principal Investigator. Patients must be willing to have a tumor biopsy if adequate archival tissue is not available (i.e., post-enrollment and prior to treatment).
3. Measurable lymph nodes or masses of at least 1.5 centimeters (cm) on baseline CT or MRI
4. Stage II, III, or IV disease as classified by the Ann Arbor Classification
5. Age greater than or equal to 18 years
6. ECOG performance status less than or equal to 2.
7. Adequate organ and marrow function as defined below unless dysfunction is felt to be secondary to lymphoma involvement as determined by the treating investigator:

   * absolute neutrophil count* >=1,000/mcL
   * hemoglobin* >= 8 g/dL (transfusions permitted to meet criteria)
   * Platelets >= 75,000/mcL (transfusions not permitted)
   * total bilirubin <= 1.5 X institutional ULN (or <= 3 X institutional ULN for patients with documented Gilberts syndrome or cholestatic obstruction or involvement by lymphoma)
   * AST(SGOT)/ALT(SGPT) <= 3 X institutional ULN (<= 5 x ULN for patients with cholestatic obstruction or involvement by lymphoma
   * Serum creatinine <= 2.0 mg/dL

   OR

   -Creatinine clearance >=40 mL/min/1.73 m2 for patients with creatinine levels above 2 mg/dL

   *RBC transfusions and use of G-CSF will be allowed in order to meet eligibility parameters.

   NOTE: In patients without bone marrow involvement, transfusions of RBCs are permitted to achieve the criterion hemoglobin of 8g/dl, but transfusions of platelets are not permitted to achieve the criterion platelet count of >75,000/mcL. In patients with bone marrow involvement, all transfusions are permissible at the discretion of the investigator.
8. Effects of acalabrutinib on the developing human fetus are unknown. For these reasons the following measures apply:

   * Individuals of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment.
   * Individuals of childbearing potential who are sexually active must agree to highly effective contraception prior to study entry, for the duration of study participation, and for at least 2 days after the last dose of acalabrutinib or 12 months after the last dose of combined chemotherapy, whichever is later. Individuals who can father children must use highly effective contraception prior to study entry, for the duration of study participation, and for 12 months after the last dose of combined chemotherapy; there is no contraception timing requirement post-last dose of acalabrutinib alone if an individual who can father children does not initiate chemotherapy on study after the acalabrutinib window.
   * Participants must not be planning to conceive or father children within the projected duration of the trial, starting with the pre-screening/screening visit through 2 days after the last dose of acalabrutinib or 12 months after the last dose of combined chemotherapy, whichever is later.

   NOTE: An individual is considered of childbearing potential, (i.e., fertile), following menarche and until becoming post-menopausal unless permanently sterile or have a congenital or acquired condition that prevents childbearing. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy at least 6 weeks before screening. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. In individuals of childbearing potential <45 years of age, a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in individuals of childbearing potential not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient The investigator or a designated associate is requested to advise the subject how to achieve highly effective birth control (failure rate of less than 1%), e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence.

   Individuals who can father children are considered to be of non-reproductive potential if they are permanently sterile due to bilateral orchiectomy.

   Highly effective methods of contraception (to be used during heterosexual activity) are defined as methods that can achieve a failure rate of <1% per year when used consistently and correctly. Such methods include:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable
   * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomy of participant or participant's partner (with medical assessment and confirmation of vasectomy surgical success)
   * Sexual abstinence (only if refraining from heterosexual intercourse during the entire period of risk associated with the study treatments)

   Hormonal contraception may be susceptible to interaction with study or other drugs, which may reduce the efficacy of the contraception method.

   Abstinence (relative to heterosexual activity) can only be used as the sole method of contraception if it is consistently employed during the entire period of risk associated with the study treatments.

   Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, and post-ovulation methods) and withdrawal are not acceptable methods of contraception.
9. Ability of patient to understand and the willingness to sign a written informed consent document.
10. Any HIV status will be included in this study; status must be confirmed prior to enrollment.

EXCLUSION CRITERIA:

1. Patients who meet histologic criteria for the following subtypes are excluded:

   * Primary DLBCL of the central nervous system (PCNSL)
   * Primary mediastinal B-cell lymphoma (PMBL)
   * Plasmablastic lymphoma
   * Intravascular large B-cell lymphoma
   * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
2. Patients who, at the discretion of the investigator, need immediate cytoreductive chemotherapy such as patients with evidence of spontaneous tumor lysis or impending organ compromise are not eligible.
3. Current or prior anti-cancer treatment for DLBCL prior to enrollment. Short course of corticosteroids (<7 days) for acute issues prior to study enrollment are permitted.
4. Major surgical procedure within 30 days of first dose of study drug. If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
5. Requires treatment with moderate or strong CYP3A inhibitors or inducers
6. Known lymphomatous involvement of the CNS
7. Pregnant individuals, or individuals who intend to become pregnant during the study are excluded from this study because of potential teratogenic effects associated with acalabrutinib, R-CHOP, and/or DA-EPOCH-R
8. The potential for all study treatments to be excreted in the milk of nursing mothers is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with acalabrutinib, nursing must be discontinued.
9. Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient at the discretion of the investigator:

   -Other malignancy that requires ongoing systemic hormonal therapy, chemotherapy, or immunotherapy.

   Uncontrolled active systemic infection
   * Any condition that requires anticoagulation with warfarin or equivalent vitamin K antagonist
   * Active bleeding, history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
   * Suspected or confirmed Progressive Multifocal Leukoencephalopathy (PML)
   * Active hepatitis C infection. NOTE: Subjects who are hepatitis C antibody positive will need to have a negative HCV PCR result before enrollment. Those with a positive PCR for hepatitis C are excluded.
   * Active hepatitis B infection. NOTE: Patients who are hepatitis B surface antigen (HbsAg) positive will be excluded from enrollment. Patients who are hepatitis B core antibody (HbcAb) positive will need to have a negative HBV PCR result before enrollment. Those with a positive PCR for hepatitis B are excluded. Those who are hepatitis B core antibody (HbcAb) positive with a negative PCR for hepatitis B will be treated with antivirals designed to prevent hepatitis B reactivation (e.g., entecavir) throughout therapy and for 12 months after therapy and have monitoring for hepatitis B reactivation with PCR.
   * History of hemorrhagic stroke or intracranial hemorrhage in preceding 6 months
   * Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification. Subjects with controlled atrial fibrillation/flutter during screening are eligible.
   * Uncontrolled autoimmune hemolytic anemia
   * Inability to swallow oral medications, or disease involve that significantly limits absorption of oral medication
   * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study.
10. Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | every 2 cycles
  Number of patients who achieve a CR, PR or SD

SECONDARY OUTCOMES:
Safety and tolerability | initiation of study drug until 30 days after last dose
  Incidence of adverse events (i.e., grade and frequency)
Progression-free survival | every 3-6 months for 5 years then yearly
  The response rate will be determined and reported along with a 95% confidence interval.
Overall survival | every 3-6 months for 5 years then yearly
  The response rate will be determined and reported along with a 95% confidence interval.
Event-free survival | every 3-6 months for 5 years then yearly
  The response rate will be determined and reported along with a 95% confidence interval.
Complete response rate | 6 cycles
  The response rate will be determined and reported along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. @@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Roschewski M, Kurtz DM, Westin JR, Lynch RC, Gopal AK, Alig SK, Sworder BJ, Cherng HJ, Kuffer C, Blair D, Brown K, Goldstein JS, Schultz A, Close S, Chabon JJ, Diehn M, Wilson WH, Alizadeh AA. Remission Assessment by Circulating Tumor DNA in Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec;43(34):3652-3661. doi: 10.1200/JCO-25-01534. Epub 2025 Aug 13. PMID 40802906
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0116.html